CLINICAL TRIAL: NCT02028962
Title: Development, Implementation and Evaluation of a Computer Tailored Program for Smoking Cessation Among Romanian Adults
Brief Title: Computer Tailored Program for Smoking Cessation Among Romanian Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Lucia Maria Lotrean, MD, PhD, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Renuntlafumat
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Tobacco Smoking
Keywords: Smoking cessation; Romanian adults
MeSH Terms: conditions — Tobacco Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Experimental): The experimental group will receive three letters with advices for smoking cessation-the first letter after the enrolment in the study, the second one one month after the first letter, the third one three months after the first letter
  Interventions: Behavioral: Lifestyle counseling
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Lifestyle counseling
  Arms: Lifestyle counseling

SUMMARY:
The research aim is the development, implementation and evaluation of the first computer tailored smoking cessation progam for Romanian adult smokers. It will be implemented among smokers from Romania aged 20-60 years. The participants will beneficiate of tailored information received in letters generated by using sophisticated computer algorithms, allowing the creation of highly individualized messages that address each individual's unique needs, motivations and beliefs related to smoking .

Program implementation will comprise of :

1. ''diagnosis'' by means of questionnaires at the individual level of characteristics that are relevant for a person's smoking behavior
2. development of the ''message library'' that contains all education messages that may be needed
3. development of an ''algorithm'', a set of decision rules that evaluates the diagnosis, selects and generates messages tailored to the specific needs of the individual user
4. generating of personalized letters for each participant
5. sending of theses personalized letters to the participants. The participants will receive three personalized letters during a period of six months after registration into the program.

The effects of the program will be evaluated with a randomized controlled trial which will assess the changes in smoking behaviour as well as smoking related attitudes, self-efficacy and quiting attempts at 6 months after the enrolment into the program.

A process evaluation will assess participants' opinion about the program.

ELIGIBILITY:
Inclusion Criteria:

* smokers (smoked in the last 7 days)who intend to quit smoking in the next 6 months

Exclusion Criteria:

* non-smokers
* smokers who do not intend to quit smoking in the next 6 months

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 640 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-08 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
abstinence from smoking in the last 7 days | baseline and 6 months after

SECONDARY OUTCOMES:
quiting attempts in the last 6 months | baseline and 6 months after
smoking related attitudes | baseline and six months after
self-eficacy in quiting smoking | baseline and 6 months after

CONTACTS AND LOCATIONS:
Overall Officials: Lucia M Lotrean, MD, PhD, Principal Investigator — Iuliu Hatieganu University of Medicine and Pharmacy, Cluj-Napoca, Romania
Locations (1):
- Iuliu Hatieganu University of Medicine and Pharmacy, Cluj-Napoca, Cluj, Romania

REFERENCES:
- See also: Related Info — http://renuntlafumat.umfcluj.ro